CLINICAL TRIAL: NCT02355444
Title: Dietary Intervention to Investigate the Effects of Blackberry-derived Polyphenols on Cardio-metabolic Risk Factors in Adults
Brief Title: Effects of Blackberry-derived Polyphenols on Cardiovascular Risk in Adults
Acronym: Cardio-Rubus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Alice Lucey, Research Fellow, University College Cork
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Cardio-rubus 13F539
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose blackberry polyphenol beverage (Experimental): Each participant will consume a blackberry beverage with high-dose blackberry polyphenols (250mL/day for 6 weeks).
  Interventions: Dietary Supplement: blackberry polyphenol enriched beverage
- Low-dose blackberry polyphenol beverage (Placebo Comparator): Each participant will consume a blackberry beverage with minimal blackberry polyphenols (250mL/day for 6 weeks).
  Interventions: Dietary Supplement: blackberry beverage with minimal polyphenol concentrations

INTERVENTIONS:
Dietary Supplement: blackberry polyphenol enriched beverage — Double-blind intervention study, cross-over design with one 250 mL bottle of high-dose blackberry polyphenol beverage per day or placebo (blackberry beverage with minimal polyphenol) in Phase one followed by cross-over in Phase two.
  Other Names: Rubus Fructicosus
  Arms: High-dose blackberry polyphenol beverage
Dietary Supplement: blackberry beverage with minimal polyphenol concentrations — Double-blind intervention study, cross-over design with one 250 mL bottle of high-dose blackberry polyphenol beverage per day or placebo (blackberry beverage with minimal polyphenol) in Phase one followed by cross-over in Phase two.
  Other Names: Rubus Fructicosus
  Arms: Low-dose blackberry polyphenol beverage

SUMMARY:
Cardiovascular disease (CVD) is the most common cause of death in Ireland, accounting for 33% of all deaths. Hypertension or elevated blood pressure, is also a significant health problem, however, it is one of the major controllable risk factors associated with CVD. While increased consumption of fruit and vegetables is associated with reduced risk of CVD, evidence is accumulating that consumption of berry fruits in particular, may promote cardiovascular health. Blackberries have a favourable nutritional profile, in that they are rich in dietary fibre, vitamins C, K and folate but low in dietary fat and kilocalories. In addition, blackberries are a rich source of antioxidants, and contain numerous phytochemicals including polyphenols. The aim of this study is to investigate the potential beneficial effects of blackberry consumption on cardiovascular health, in particular, effects on blood pressure.

DETAILED DESCRIPTION:
Dietary factors play a significant role in the prevention and/or treatment of hypertension and significant efforts are being put in to the development of functional foods with antihypertensive activity. Blackberries and their intrinsic polyphenols, consumed as part of a healthy diet, may be of functional interest in both the treatment and prevention of hypertension and dyslipidaemia. The Cardio-Rubus study presents healthy adults with an opportunity to participate in a human nutrition study that will assist in identifying biological effects of blackberry-derived components establishing further the value of berries as a nutritious, health conducive food.

It is proposed to carry out a crossover, randomized double-blind 18-week supplementation study in 100 men and women aged 45-70 years with a systolic blood pressure of 130-149 mmHg but who are otherwise in good health. The proposed sample size is based on systolic blood pressure data derived from baseline values of 700 adults who participated in RCTs that we have conducted at UCC over the last 6-7 years. The calculation for sample size is based on observational data of systolic blood pressure in older pre-hypertensive adults, which showed a mean (SD) SBP of 135 (3) mmHg. The proposed study is powered to detect a mean drop of 2 mmHg systolic blood pressure at 85% power and with a significance level of 5%. The calculations support the recruitment of 100 participants in total (n = 41 per group, rounded up to 50 to account for a 20% attrition rate).

Potential study participants will be recruited by researchers at the School of Food & Nutritional Sciences and all study visits will take place at the Human Nutrition Studies Unit, UCC. In addition to the provision of written information, the study protocol will be clearly and comprehensively discussed with each potential participant prior to enrollment and their provision of informed written consent. Participants will initially complete a 2-week run in period which involves refraining from the consumption of specified foods items (predominantly berries and other fruits) until the end of the study. Each participant will be randomly assigned to receive one of two beverages (either a high dose or low dose blackberry polyphenol enriched beverage) for a period of 6-weeks (study phase 1) and then after a 2-week wash-out, the participant will receive the opposite treatment to that which was provided during study phase 1 for the next 6-weeks (study phase 2). After completion of study phase 2 there will be a 2-week wash-out followed by a final visit to UCC. Thus, after screening and enrolment on to the study, there will be a further 5 visits to UCC (at the baseline and endpoint of each study phase and at the end of the final washout phase). All 5 visits will be fasting morning visits where the nurse will take a small blood sample which will be analysed for blood lipids, fasting glucose and biomarkers of endothelial function. Brachial and central blood pressure will be measured as well as an assessment of arterial stiffness by pulse wave velocity analysis. Body weight, BMI and waist circumference will also be measured. Each participant's body composition (% body fat & lean mass) will be assessed by DXA scan.

All information collected is strictly confidential. Samples and questionnaires will be labelled with a unique identifying code, and participant's names will not be used at any stage during data collection, database construction or data analysis. Data will be archived by the principal investigator. In any publications or other documents, participants will not be identified by name or code numbers. Group summary data will be presented in place of individual data, further ensuring confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adult Caucasian men and women (ratio men: women, 70:30)
* Good general health
* Systolic blood pressure: 130 - 149 mmHg
* Body mass index (BMI): 25.0 - 35.0 kg/m2
* Signed consent form

Exclusion Criteria:

* Current smokers
* Diagnosed hypertension
* History of cardiovascular events such as stroke, myocardial infarction or peripheral vascular disease
* Diagnosed medical illness including diabetes mellitus (Types 1 & 2), chronic kidney disease and gastro-intestinal diseases
* Medications that may affect any of the study outcome measures: anti-hypertensive medications and lipid lowering therapies e.g. statins.
* Suspected hypersensitivity or allergy to berries.
* Intolerance for aspirin or salicylate acid.
* Current consumption of nutraceuticals, botanical extracts or other polyphenol-rich supplements.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 42 days
  A change between baseline blood pressure and endpoint blood pressure within the intervention group versus the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Mairead Kiely, PhD, Principal Investigator — School of Food & Nutritional Sciences, University College Cork.
Locations (1):
- Human Nutrition Studies Unit, School of Food & Nutritional Sciences, UCC, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided